CLINICAL TRIAL: NCT00600626
Title: Comparison of Basal Bolus Treatment With Insulin Aspart Including Insulin NPH and Biphasic Insulin Aspart in Type 2 Diabetes Mellitus
Brief Title: Basal Bolus of Insulin Aspart Including Insulin NPH and Biphasic Insulin Aspart in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1486
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: insulin NPH
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe and Asia. The aim of this trial is to compare basal bolus treatment with insulin aspart and insulin NPH to biphasic insulin aspart treatment on blood glucose control in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with human insulin or insulin analogues for at least 3 months, with or without combination with OADs
* HbA1c between 8.0-10.5%
* Body mass index (BMI) below 35.0 kg/m2
* Able and willing to perform self-monitoring of blood glucose

Exclusion Criteria:

* Total daily insulin dose of 1.80 IU/kg or more
* Known or suspected allergy to trial product or related products
* Pregnancy, breast-feeding, the intention to become pregnant or judged not to be using adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2004-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 4 months of treatment

SECONDARY OUTCOMES:
8-point blood glucose profile
incidence of hypoglycaemic episodes
safety profiles
changes in body weight and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (52):
- Novo Nordisk Investigational Site, Zagreb, Croatia
- France (4):
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (8):
  - Novo Nordisk Investigational Site, Bad Heilbrunn
  - Novo Nordisk Investigational Site, Neuss
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Schaafheim
  - Novo Nordisk Investigational Site, Schwedt
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wiesbaden
  - Novo Nordisk Investigational Site, Würzburg
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Malaysia (2):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
- Netherlands (4):
  - Novo Nordisk Investigational Site, Beverwijk
  - Novo Nordisk Investigational Site, Delft
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Rotterdam
- Poland (5):
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Romania (4):
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Constanța
  - Novo Nordisk Investigational Site, Iași
  - Novo Nordisk Investigational Site, Timișoara
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Singapore, Singapore
- Spain (6):
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Orihuela
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valladolid
- Sweden (6):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Mölndal
  - Novo Nordisk Investigational Site, Uppsala
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Brighton
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, York

REFERENCES:
- [Result] Ligthelm RJ, Mouritzen U, Lynggaard H, Landin-Olsson M, Fox C, le Devehat C, Romero E, Liebl A. Biphasic insulin aspart given thrice daily is as efficacious as a basal-bolus insulin regimen with four daily injections: a randomised open-label parallel group four months comparison in patients with type 2 diabetes. Exp Clin Endocrinol Diabetes. 2006 Oct;114(9):511-9. doi: 10.1055/s-2006-924424. PMID 17115349
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com